CLINICAL TRIAL: NCT01310400
Title: Observer-blind, Randomized, Controlled Study to Determine the Immunogenicity and Safety of a Two-dose Regimen of Virosomal Subunit Influenza Vaccine Inflexal V in Healthy Young Children (≥6 Months to ≤35 Months) in Comparison With the Subunit Influenza Vaccine Agrippal
Brief Title: Comparison of the Efficacy of Inflexal V With a Commercially Available Influenza Vaccine in Young Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TG0826INF
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2013-08

CONDITIONS: Influenza
Keywords: Influenza; Virus; Vaccination; Immunisation
MeSH Terms: conditions — Influenza, Human; Virus Diseases | interventions — Inflexal V

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Inflexal 0.5 mL (Experimental)
  Interventions: Biological: Inflexal V
- Inflexal 0.25 mL (Experimental)
  Interventions: Biological: Inflexal V
- Agrippal 0.25 mL (Experimental)
  Interventions: Biological: Agrippal

INTERVENTIONS:
Biological: Inflexal V — Inflexal V influenza vaccine, formulated for the WHO requirements of the 2009-2010 season, containing per 0.5 mL dose:
  * 15 µg hemagglutinin (HA) antigen of A/Brisbane/59/2007 (H1N1)-like virus
  * 15 µg HA antigen of A/Brisbane/10/2007 (H3N2)-like virus
  * 15 µg HA antigen of B/Brisbane/60/2008-like virus
  Dose: intramuscular administration (M. deltoideus) of a single dose of 0.5 mL on Days 0 and 28
  Arms: Inflexal 0.5 mL
Biological: Inflexal V — Inflexal V influenza vaccine, formulated for the WHO requirements of the 2009-2010 season, containing per 0.5 mL dose:
  * 15 µg HA antigen of A/Brisbane/59/2007 (H1N1)-like virus
  * 15 µg HA antigen of A/Brisbane/10/2007 (H3N2)-like virus
  * 15 µg HA antigen of B/Brisbane/60/2008-like virus
  Dose: intramuscular administration (M. deltoideus) of a single dose of 0.25 mL on Days 0 and 28
  Arms: Inflexal 0.25 mL
Biological: Agrippal — Agrippal influenza vaccine
  Dose: intramuscular administration (M. deltoideus) of a single dose of 0.25 mL on Days 0 and 28
  Arms: Agrippal 0.25 mL

SUMMARY:
A study to assess whether the Northern Hemisphere 2009/2010 season influenza vaccine Inflexal V is as immunogenic as a locally sourced competitor vaccine in young children.

ELIGIBILITY:
Inclusion Criteria:

* ≥6months to ≤35 months-old healthy children (male or female) born at term after normal pregnancy
* Recording of medical history and physical examination reveal no abnormality
* The parent/legal guardian of the participating child must sign the written informed consent and agree to provide a blood sample taken from the child pre- and post-immunization

Exclusion criteria:

* Hypersensitivity to eggs, chicken proteins, polymyxin B, neomycin or any component of the vaccine
* Previous vaccination against influenza
* At time of enrollment, presentation of clinical symptoms of active infection and/or body temperature ≥38°C
* Confirmation or suspicion of immunosuppressed status (including cancer), or confirmation of immunodeficiency disease (congenital or acquired including HIV)
* Medical treatment (>2 weeks) with immune suppressant or immune modulating drugs including systemic steroids during the last 3 months before immunization or at present, as follows: long-term oral prednisone or other equivalent steroid: ≥0.5mg/kg/day (note: administration of local or inhaled steroids before or during the study is allowed)
* Treatment with immunoglobulins or blood products during the last 3 months before immunization or such treatment scheduled during the study
* Participation in other clinical trials during the last 3 months before immunization or intention to participate during this study period
* At present or during the last 6 months before immunization: radiotherapy or treatment with cytotoxic drugs
* Other vaccination with a killed vaccine within 14 days before immunization or with an attenuated vaccine within 28 days before immunization (note: after subject inclusion vaccines of the immunization program for children are allowed upon the physician's discretion. However, immunization on the same day must be avoided)
* Family history of Guillain-Barré Syndrome
* Severe congenital deficiency or disease
* Antecedent of neurological disease or epileptic attack
* Severe cardiopulmonary disease with possibility to influence the study result
* Disturbance of coagulation or under anticoagulant treatment, likely to be contraindicated to i.m. injection
* Suspected non-compliance

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1356 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rongcheng Li, MD, Principal Investigator — Guangxi Zhuang Autonomous Region CDC
Locations (1):
- Guangxi Zhuang Autonomous Region CDC, Nanning, Guangxi, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Inflexal V 0.5 mL; Inflexal V 0.25 mL; Agrippal 0.25 mL: Subjects received 2 doses: 1st dose on Day 0, 2nd dose on Day 28
Period: Overall Study
Arm/Group | Inflexal V 0.5 mL | Inflexal V 0.25 mL | Agrippal 0.25 mL
Started | 452 | 452 | 452
Completed | 424 | 420 | 422
Not Completed | 28 | 32 | 30

BASELINE CHARACTERISTICS:
Groups:
- Inflexal V 0.5 mL: The safety data are shown for the safety population (N = 452 for this group).
- Inflexal V 0.25 mL; Agrippal 0.25 mL: The safety data are shown for the safety population (N = 451 for this group).
- Total: Total of all reporting groups
Arm/Group | Inflexal V 0.5 mL | Inflexal V 0.25 mL | Agrippal 0.25 mL | Total
Number analyzed (Participants) | 452 | 451 | 451 | 1354
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 452 | 451 | 451 | 1354
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.8 (0.7) | 1.8 (0.7) | 1.8 (0.7) | 1.8 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 227 | 215 | 206 | 648
  Male | 225 | 236 | 245 | 706
Region of Enrollment [Number; unit: participants]
  China | 452 | 451 | 451 | 1354

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity, Assessed by the Haemagglutination (HI) Test
Description: Seroconversion rate post-immunization. Seroconversion is defined as a post-vaccination titer of ≥1:40 for those with a pre-vaccination HI titer of <1:10 and as ≥ four-fold increase in HI titer for those with a pre-vaccination HI titer of ≥1:10.
Time Frame: 3 weeks after the 2nd vaccination
Population: According-to-protocol population: subjects who received both doses of influenza vaccine, with available pre- and post-vaccination titers and without major protocol violations
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Inflexal V 0.5 mL: The immunogenicity results are shown for the per-protocol population (N = 423 for this group).
- Inflexal V 0.25 mL: The immunogenicity results are shown for the per-protocol population (N = 380 for this group).
- Agrippal 0.25 mL: The immunogenicity results are shown for the per-protocol population (N = 384 for this group).
Arm/Group | Inflexal V 0.5 mL | Inflexal V 0.25 mL | Agrippal 0.25 mL
Number analyzed (Participants) | 423 | 380 | 384
percentage of participants
  Percentage of subjects seroconverted: A/H1N1 | 97.2 [95.1 to 98.5] | 89.7 [86.2 to 92.6] | 92.7 [89.6 to 95.1]
  Percentage of subjects seroconverted: A/H3N2 | 90.5 [87.4 to 93.2] | 83.4 [79.3 to 87.0] | 82.6 [78.4 to 86.2]
  Percentage of subjects seroconverted: B-strain | 57.5 [52.6 to 62.2] | 47.9 [42.8 to 53.1] | 37.2 [32.4 to 42.3]
Statistical Analysis 1: Comparison: Inflexal V 0.5 mL vs Agrippal 0.25 mL; This statistical anaylsis evaluated the non-inferiority of 0.5 mL Inflexal V vs. 0.25 mL Agrippal for the A/H1N1 strain; Test type: Non-Inferiority or Equivalence — This study evaluated the non-inferiority of 0.5 mL Inflexal V and 0.25 mL Inflexal V in comparison to 0.25 mL Agrippal. Seroconversion rate was the primary endpoint. The difference in seroconversion rates between each Inflexal V and the control group was used for the evaluation of non-inferiority. If the lower limit of the 95% CI of this difference was greater than -10% for all 3 strains, the Inflexal V group was considered non-inferior to the control group; p = 0.0036, Chi-squared — The significance level α = 0.05 (one-sided) was adjusted to α = 0.025 (one-sided) for the primary endpoint; Difference in seroconversion rates = 4.5, 95% CI 2-sided [1.4 to 7.5]
Statistical Analysis 2: Comparison: Inflexal V 0.25 mL vs Agrippal 0.25 mL; This statistical anaylsis evaluated the non-inferiority of 0.25 mL Inflexal V vs. 0.25 mL Agrippal for the A/H1N1 strain; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.1465, Chi-squared — The significance level α = 0.05 (one-sided) was adjusted to α = 0.025 (one-sided) for the primary endpoint; Difference in seroconversion rates = -3.0, 95% CI 2-sided [-7.0 to 1.0]
Statistical Analysis 3: Comparison: Inflexal V 0.5 mL vs Agrippal 0.25 mL; This statistical anaylsis evaluated the non-inferiority of 0.5 mL Inflexal V vs. 0.25 mL Agrippal for the A/H3N2 strain; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Chi-squared — The significance level α = 0.05 (one-sided) was adjusted to α = 0.025 (one-sided) for the primary endpoint; Difference in seroconversion rates = 8.0, 95% CI 2-sided [3.3 to 12.7]
Statistical Analysis 4: Comparison: Inflexal V 0.25 mL vs Agrippal 0.25 mL; This statistical anaylsis evaluated the non-inferiority of 0.25 mL Inflexal V vs. 0.25 mL Agrippal for the A/H3N2 strain; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.7493, Chi-squared — The significance level α = 0.05 (one-sided) was adjusted to α = 0.025 (one-sided) for the primary endpoint; Difference in seroconversion rates = 0.9, 95% CI 2-sided [-4.5 to 6.2]
Statistical Analysis 5: Comparison: Inflexal V 0.5 mL vs Agrippal 0.25 mL; This statistical anaylsis evaluated the non-inferiority of 0.5 mL Inflexal V vs. 0.25 mL Agrippal for the B-strain; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0000, Chi-squared — The significance level α = 0.05 (one-sided) was adjusted to α = 0.025 (one-sided) for the primary endpoint; Difference in seroconversion rates = 20.2, 95% CI 2-sided [13.5 to 27.0]
Statistical Analysis 6: Comparison: Inflexal V 0.25 mL vs Agrippal 0.25 mL; This statistical anaylsis evaluated the non-inferiority of 0.25 mL Inflexal V vs. 0.25 mL Agrippal for the B-strain; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0029, Chi-squared — The significance level α = 0.05 (one-sided) was adjusted to α = 0.025 (one-sided) for the primary endpoint; Difference in seroconversion rates = 10.7, 95% CI 2-sided [3.7 to 17.6]

2. Secondary Outcome: Fold Increase in Geometric Mean Titer (GMT)
Description: GMT-fold increase - calculated as the GMT on Day 49 divided by the baseline GMT value
Time Frame: 3 weeks after the 2nd vaccination
Measure: Number; unit: Fold (ratio)
Arm/Group | Inflexal V 0.5 mL | Inflexal V 0.25 mL | Agrippal 0.25 mL
Number analyzed (Participants) | 423 | 380 | 384
Fold (ratio)
  GMT fold increase from baseline: A/H1N1 | 36.6 | 25.9 | 25.4
  GMT fold increase from baseline: A/H3N2 | 72.5 | 48.8 | 54.2
  GMT fold increase from baseline: B-strain | 9.2 | 7.0 | 5.3

3. Secondary Outcome: Seroprotection
Description: Seroprotection rate, defined as a post-vaccination HI titer of 1:40.
Time Frame: 3 weeks after the 2nd vaccination
Measure: Number (95% Confidence Interval); unit: percentage seroprotected subjects
Arm/Group | Inflexal V 0.5 mL | Inflexal V 0.25 mL | Agrippal 0.25 mL
Number analyzed (Participants) | 423 | 380 | 384
percentage seroprotected subjects
  Percentage of subjects seroprotected: A/H1N1 | 97.6 [95.7 to 98.9] | 92.1 [88.9 to 94.6] | 93.2 [90.2 to 95.5]
  Percentage of subjects seroprotected: A/H3N2 | 91.3 [88.1 to 93.8] | 84.5 [80.4 to 88.0] | 82.8 [78.7 to 86.5]
  Percentage of subjects seroprotected: B-strain | 60.3 [55.4 to 65.0] | 51.3 [46.2 to 56.5] | 39.6 [34.7 to 44.7]

4. Secondary Outcome: Safety: Incidence of Solicited and Unsolicited Adverse Events
Description: Safety assessements were made by the investigator at baseline and on Days 28 and 49, as well as by the subjects themselves (in Subjects Diaries) for the 4-day period following each vaccination.
Time Frame: Solicited AEs: Days 1-4 and 28-31, and Days 28 and 49; unsolicited AEs: until study end
Measure: Number; unit: percentage of subjects with AEs
Arm/Group | Inflexal V 0.5 mL | Inflexal V 0.25 mL | Agrippal 0.25 mL
Number analyzed (Participants) | 452 | 451 | 451
percentage of subjects with AEs
  Subjects with at least one AE | 38.5 | 33.0 | 35.7
  Subjects with at least one solicited AE | 32.3 | 29.1 | 29.5
  Subjects with at least one unsolicited AE | 12.6 | 8.2 | 12.2

ADVERSE EVENTS:
Arm/Group | Inflexal V 0.5 mL | Inflexal V 0.25 mL | Agrippal 0.25 mL
Serious Adverse Events (participants affected / at risk) | 0/452 | 1/451 | 1/451
Other Adverse Events (participants affected / at risk) | 57/452 | 37/451 | 55/451
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inflexal V 0.5 mL (N=452) | Inflexal V 0.25 mL (N=451) | Agrippal 0.25 mL (N=451)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inflexal V 0.5 mL (N=452) | Inflexal V 0.25 mL (N=451) | Agrippal 0.25 mL (N=451)
Diarrhea (Gastrointestinal disorders) | 11 (11) | 9 (9) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 11 (11) | 23 (23)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 9 (9) | 17 (17)
Vomiting (Gastrointestinal disorders) | 16 (16) | 11 (11) | 12 (12)
Pyrexia (body temp. >=38°C) (General disorders) | 43 (43) | 31 (31) | 38 (38)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release. A time period for this review is not specified in the study protocol.